CLINICAL TRIAL: NCT06727734
Title: Levonorgestrel-piroxicam Combination Versus Ulipristal Acetate for Emergency Contraception: a Randomised Double-blind Controlled Trial
Brief Title: Levonorgestrel-piroxicam Versus Ulipristal Acetate for Emergency Contraception
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Family Planning Association of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 24-054
Record Dates: First submitted 2024-11-28; First posted 2024-12-11 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Contraception
MeSH Terms: interventions — Levonorgestrel; Piroxicam; ulipristal acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LNG-piroxicam (Experimental): Levonorgestrel-piroxicam combination
  Interventions: Drug: Levonorgestrel; Drug: Piroxicam; Drug: Placebo - UPA
- UPA (Active Comparator): Ulipristal only
  Interventions: Drug: Ulipristal Acetate; Drug: Placebo - LNG; Drug: Placebo - Piroxicam

INTERVENTIONS:
Drug: Levonorgestrel — Levonorgestrel 1.5 mg
  Other Names: Anlitin
  Arms: LNG-piroxicam
Drug: Piroxicam — Piroxicam 40 mg
  Other Names: CP-Pirox
  Arms: LNG-piroxicam
Drug: Ulipristal Acetate — Ulipristal 30 mg
  Other Names: Ella
  Arms: UPA
Drug: Placebo - LNG — Placebo of levonorgestrel
  Arms: UPA
Drug: Placebo - Piroxicam — Placebo of piroxicam
  Arms: UPA
Drug: Placebo - UPA — Placebo of ulipristal acetate
  Arms: LNG-piroxicam

SUMMARY:
The goal of this clinical trial is to compare the failure rate of the levonorgestrel (LNG)-piroxicam combination regimen versus ulipristal acetate (UPA) as emergency contraception (EC). The main questions it aims to answer are:

1. whether the LNG-piroxicam combination regimen has a lower failure rate than UPA for EC;
2. whether the LNG-piroxicam combination regimen has a higher percentage of pregnancies prevented than UPA for EC
3. whether there is any difference in the change in the subsequent menstrual cycle and adverse effect profile between the two regimens

Participants will:

1. Take a single dose of either (i) LNG 1.5 mg plus piroxicam 40 mg and a placebo tablet resembling UPA, or (ii) UPA 30 mg plus placebo tablets resembling LNG and piroxicam.
2. Have a blood test for serum LH, oestradiol an progesterone.
3. Keep a diary of their vaginal bleeding episodes, adverse effects symptoms, any further acts of intercourse and the type of contraception used.
4. Have a follow-up either in person by phone about 1-2 weeks after the next expected menstruation.
5. If normal menstrual bleeding has not occurred by that time, a pregnancy test will be carried out.

DETAILED DESCRIPTION:
Participating women will be randomised to either the LNG-piroxicam group or UPA group in 1:1 ratio according to a computer-generated randomisation list in varying blocks. Serially numbered vouchers bearing the drug code in sealed envelopes will be prepared, according to which the study medication will be prepacked by another research nurse not directly involved in patient contact in this study. The subjects, clinicians and research staff with patient contact will be blinded to the group assignment. The codes for the treatment groups will only be revealed to the investigators after completion of the whole study and statistical analyses.

Baseline assessment of subjects:

* Medical and menstrual history will be taken.
* Measurement of body height, weight and blood pressure.
* Pregnancy test
* Measurement of serum LH, oestradiol and progesterone to classify the subject as pre-ovulatory versus post-ovulatory. The serum hormonal levels will be used to estimate the phase of the menstrual cycle at the time of presentation in relation to the day of ovulation.

Treatment:

The recruited subjects will receive the assigned study medications under direct supervision. Those in the LNG-piroxicam group will receive piroxicam 40 mg, LNG 1.5 mg and a placebo pill resembling UPA. Those in the UPA group will receive UPA 30 mg and placebo pills resembling LNG and piroxicam respectively. They will be given a diary chart to record vaginal spotting and bleeding, possible side effects and further acts of intercourse, if any, and the contraceptive method used.

Follow-up:

A follow-up (either in person or by phone as pre-agreed at recruitment) will be arranged by the research nurse about 1-2 weeks after the next expected menstruation (this is incorporated into her routine clinic follow-up). Information collected at the follow-up visit will include side effects and vaginal bleeding/spotting marked by the subject on her diary card, time of onset, duration and amount of menstrual bleeding, any further acts of intercourse and the type of contraception used. If normal menstrual bleeding has not occurred by that time, a pregnancy test will be carried out, and a positive result denotes treatment failure and the woman will be counselled accordingly. Those deciding to continue with pregnancy will be referred for antenatal care. An additional research follow-up will be arranged post-delivery to record any antenatal, postnatal and neonatal complications. If the woman opts for terminating the pregnancy, she will be referred to the appropriate services. If the woman misses the appointment and does not contact the clinic, the researchers will reach her by phone (either voice call or text messaging) as soon as possible after the missed visit.

ELIGIBILITY:
Inclusion Criteria:

1. women aged 18-45 years;
2. requesting an oral EC within 120 hours of a single or the first act of unprotected intercourse in the current menstrual cycle;
3. available for follow-up over the next 6 weeks.

Exclusion Criteria:

1. post-abortion or postpartum and period have not yet returned,
2. being on the following drugs currently: anticoagulants, cyclosporine, tacrolimus, corticosteroids, lithium, serotonin reuptake inhibitors (SSRIs), quinolones
3. having unprotected intercourse in this cycle more than 120 hours before attending the clinic,
4. being found pregnant at the time of presentation,
5. breastfeeding,
6. having been sterilized (or partner having been sterilized) or having intrauterine contraceptive device in-situ,
7. uncertain about the date of the last menstrual period,
8. having used a hormonal contraceptive (including EC), progestogen-containing medication or NSAID in the recent one week,
9. having history of asthma, urticaria or other allergic reactions to piroxicam, aspirin or other NSAIDs,
10. having history of ischaemic heart disease, heart failure, hypertension, cerebrovascular disease or kidney failure requiring dialysis
11. having history of peptic ulcer disease and/or gastrointestinal bleeding.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological gender
Enrollment: 980 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | 1 month
  Percentage of women having positive hCG test within one month

SECONDARY OUTCOMES:
Percentage of pregnancies prevented | 1 month
  Percentage of pregnancies (based on published theoretical model) that are prevented in the treatment group
Change in bleeding pattern | 1 month
  Percentage of women experiencing changes to menstrual bleeding pattern within one month
Adverse effects | 1 month
  Percentage of women experiencing other adverse effects within one month

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Hang Wun Li, MD, FRCOG, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: From commencement of the study till 3 years after study completion
Access Criteria: Upon reasonably request made to the principal investigator